CLINICAL TRIAL: NCT00191490
Title: A Multicenter Randomized Phase II Study Evaluating the Feasibility and Activity of Two Different Combinations of Docetaxel (RP56976, TAXOTERE *) and Gemcitabine and of Cisplatin/Gemcitabine Followed by Docetaxel as First Line Therapy for Locally Advanced Unresectable or Metastatic Non Small Cell Lung Cancer
Brief Title: A Randomized Study Evaluating the Feasibility and Activity of Three Different Combination With Gemcitabine as First Line Therapy for Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Aventis Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6549; B9E-IT-JHSC
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Docetaxel; Cisplatin

INTERVENTIONS:
Drug: Gemcitabine
Drug: docetaxel
Drug: cisplatin

SUMMARY:
Phase II study that will evaluate the activity of gemcitabine as intravesical therapy on the marker lesion in superficial bladder carcinoma at intermediate risk. Primary objective is the evaluation of the pathological complete response after 8 instillation of gemcitabine. 46 patients are requested.

ELIGIBILITY:
Inclusion criteria

* Histologically or cytologically confirmed diagnosis of NSCLC
* Patients must have a locoregionally advanced unresectable non metastatic NSCLC Stage IIIB (only N3 supraclavicular or T4 for pleural effusion) or Stage IV according to the revised International Staging System
* Patients must have at least one measurable lesion
* WHO Performance Status 0 or 1
* Adequate Organ Function

Exclusion criteria:

* Prior systemic chemotherapy or immunotherapy including neoadjuvant or adjuvant treatments
* Prior radiotherapy for NSCLC
* Patients with symptomatic brain metastases or with leptomeningeal disease. However, patients with symptomatic brain metastases who become asymptomatic under corticosteroids treatment can enter the study
* Current peripheral neuropathy NCI grade 2

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162
Dates: Start 2002-07; Study Completion 2005-05

PRIMARY OUTCOMES:
To assess the antitumour activity as measured by response rate in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) of two different combinations of docetaxel and gemcitabine and of a sequential treatment of
cisplatin /gemcitabine

SECONDARY OUTCOMES:
To determine time to progression, duration of response, time to treatment failure, and overall survival in each group.
To evaluate changes from baseline in the Lung Cancer Symptom Scale of patients in each treatment arm

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) Monday-Friday 9am-5pm Eastern time (UTC/GMT - 5 hours, EST), Study Chair — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, please call 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559), Monday-Friday, 9:00 am to 5:00 pm Eastern time (UTC/GMT - 5 hours, EST) or speak with your physician, Sesto Fiorentino, Florence, Italy